CLINICAL TRIAL: NCT06216574
Title: Optimizing Psychosocial Intervention for Breast Cancer-Related Sexual Morbidity:The Sexual Health and Intimacy Education (SHINE) Trial
Brief Title: Developing an Internet-Delivered Sexual Health Program for Breast Cancer Survivors, SHINE Trial
Acronym: SHINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00104518; NCI-2023-06866 (Registry Identifier: NCI CTRP); WF-2202 (Other: Wake Forest NCORP Research Base); R37CA269776 (NIH)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; sexual health; factorial MOST design
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Factorial trial using the multiphase optimization strategy (MOST) framework, in which participants will be randomized to one of 16 conditions (2^4) to receive access to a combination of one to four SHINE components.
Who Masked: Investigator
Masking Description: Local NCORP site staff and study investigators will be blinded to the treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- SHINE 1 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - 45 minutes, 4) Intimacy - 45 minutes Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 2 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - 45 minutes, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Interventions: Other: Internet-based Intervention
- SHINE 3 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - NONE, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 4 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - NONE, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Interventions: Other: Internet-based Intervention
- SHINE 5 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - 45 minutes, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 6 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - 45 minutes, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Interventions: Other: Internet-based Intervention
- SHINE 7 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - NONE, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 8 (Experimental): SHINE components assigned: 1) Psycho-education (Enhanced) - 45 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - NONE, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy. Enhanced version is tailored, interactive instruction and recommendations for over-the-counter products and aids.
  Interventions: Other: Internet-based Intervention
- SHINE 9 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - 45 minutes, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 10 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - 45 minutes, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Interventions: Other: Internet-based Intervention
- SHINE 11 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - NONE, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 12 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - 45 minutes, 3) Communication with Partner - NONE, 4) Intimacy -NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Communication with the clinician reviews clinical terminology to describe physical symptoms of sexual concern and potential scripts for discussion with an appropriate clinician.
  Interventions: Other: Internet-based Intervention
- SHINE 13 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - 45 minutes, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 14 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - 45 minutes, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Communication with partner provides effective models and exercises to practice clear communication regarding sexual concerns with partner.
  Interventions: Other: Internet-based Intervention
- SHINE 15 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - NONE, 4) Intimacy - 45 minutes.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Intimacy module provides strategies for increasing non-sexual intimacy, reconsidering sexual scripts, and focus exercises.
  Interventions: Other: Internet-based Intervention
- SHINE 16 (Experimental): SHINE components assigned: 1) Psycho-education (Standard) - 20 minutes, 2) Communication with Clinician - NONE, 3) Communication with Partner - NONE, 4) Intimacy - NONE.
  Each component is a single lesson accessed at participant's convenience and may be repeated.
  Standard psycho-education has content on effects of cancer on sexual function, self-image, and relationships, managing sexual concerns, and basic sexual anatomy.
  Interventions: Other: Internet-based Intervention

INTERVENTIONS:
Other: Internet-based Intervention — Receive access to SHINE modules

SUMMARY:
The goal of this clinical trial is to develop an effective internet-delivered program to help breast cancer survivors manage cancer-related sexual concerns.

This study is being done to find out if the study approach is better or worse than the usual approach to helping breast cancer survivors manage cancer-related sexual concerns. The usual approach is defined as care most cancer survivors get for their cancer-related sexual concerns.

Participants will complete a questionnaire and if they qualify, they will be assigned to one of sixteen groups of participants. Groups will get access to various kinds of help through an Internet-delivered program called SHINE, which was designed and is run by researchers at the University of Virginia Center for Behavioral Health and Technology. All groups will get access to education about sexual health after cancer: either a standard education website or an enhanced education web program. Groups may also receive up to three additional web programs on: talking to your clinicians about sexual concerns, and/or talking to your partner about sexual concerns, and/or increasing intimacy. Participants are asked to complete the SHINE program within 12 weeks.

After participants finish this 12-week period, the study team will ask them to complete a questionnaire to check in with the participant. The participant will be asked one additional time 12 weeks later to complete another questionnaire to see how the participant is doing. A participant will be in the study for 24 weeks.

DETAILED DESCRIPTION:
This study has sixteen study groups with about twenty people in each group. Different groups receive different combinations of help. Participants will receive a certain combination of these four different Cores to make up their SHINE program. A Core is equal to one 20-45-minute lesson. Participants will receive access to all assigned Cores at one time. Participants can complete them at their own pace, as the SHINE program allows them to return where they left off. The four Cores are described below:

* Education Core: A one-time education about sexual health after breast cancer by either a traditional webpage or by a web-based program. In the traditional webpage, a participant can read and review the information at their own pace. In the web-based program, a participant can also read and review the information at their own pace, and the information will be presented with interactive activities and email reminders. This one-time lesson should take the participant 20-45 minutes to complete.
* Talking with a Clinicians Core: A participant may receive access to a web-based program about how to talk with their health care team about their sexual concerns. A participant can use this program at their own pace, and it will have information, activities, and email reminders. This one-time lesson should take a participant approximately 45 minutes to complete.
* Talking with a Partner Core: A participant may receive access to a web-based program about how to talk with their partner about their sexual concerns. A participant can use this program at their own pace, and it will have information, activities, and email reminders. This one-time lesson should take a participant approximately 45 minutes to complete.
* Intimacy Enhancement Core: A participant may receive access to a web-based program about how to increase their physical and emotional closeness with their partner. A participant can use this program at their own pace, and it will have information, activities, and email reminders. This one-time lesson should take the participant approximately 45 minutes to complete.

Before you begin the study, your medical team will review your medical record. This helps your medical team decide if it is safe for you to take part in the study. If you join the study, you will have the usual care you would get even if you were not in the study.

If you choose to take part in this study, you will be asked to fill out forms with questions about your sexual concerns, function, symptoms, and experiences, as well as relationship satisfaction and intimacy. In addition, you will be asked about your communication about sexual concerns with your medical team and partner. Finally, you will be asked for your thoughts about the SHINE program, and a little about your demographics, distress, daily lifestyle, physical activity, and tobacco use. Researchers will use this information to determine what combination of kinds of help delivered by the internet is best for breast cancer patients to better understand and address their sexual concerns.

Participants will be asked to fill out questionnaires electronically from a link that is emailed to them three separate times during the study:

* After a participant consents, before they can be randomized to a study group.
* Approximately 12 weeks after the participant completes the first questionnaire.
* Approximately 24 weeks after the participant completes the first questionnaire.

Each questionnaire will take about 40 to 45 minutes to complete. Participants may skip any question for any reason.

ELIGIBILITY:
Inclusion Criteria:

* History of Stage 0-III breast cancer diagnosis. History of non-breast malignancies are permitted.
* ≥12 weeks following last primary cancer treatment. For this protocol, primary cancer treatments are defined as chemotherapy, cytotoxic antibody-drug conjugates, checkpoint inhibitors, radiation, and surgical procedures intended to remove malignant tissue. Ongoing adjuvant endocrine therapy (e.g., tamoxifen, aromatase inhibitors), adjuvant cdk 4/6-inhibitors (e.g., abemaciclib), HER2-based Monoclonal antibody therapy (e.g., trastuzumab, pertuzumab), HER2 targeted Tyrosine Kinase inhibitors (e.g., neratinib), and/or pending breast reconstructive surgery are allowed. (There is no upper limit on time since treatment.)
* Age ≥ 18 years at the time of study enrollment

SELF-REPORTED ELIGIBILITY SCREENER INCLUSION

* female
* Currently in an intimate relationship, as reported on the Patient-Reported Outcomes Measurement Information System Sexual Function and Satisfaction (PROMIS SexFS) screener (this relationship may be with an individual of any sex)
* Endorse being at least "somewhat" bothered by >=1 of the following during the last 30 days: (lack of) interest in sexual activity, vaginal dryness, pain during sexual activity, or (in)ability to orgasm, as reported on the PROMIS SexFS Bother Regarding Sexual Function screener
* Endorse that ≥ 1 of the bothersome sexual symptoms, from the PROMIS SexFS Bother Regarding Sexual Function screener is related to their breast cancer
* Has a working email address (or willing to create one) and receive emails from the study

Exclusion Criteria:

* Planned cancer treatment for residual, progressive, or recurrent disease within the 24 weeks following enrollment (defined as chemotherapy, cytotoxic antibody-drug conjugates, checkpoint inhibitors, radiation, and/or surgical procedures intended to remove malignant tissue). Ongoing adjuvant endocrine therapy (e.g., tamoxifen, aromatase inhibitors), adjuvant cdk 4/6-inhibitors (e.g., abemaciclib), HER2-based Monoclonal antibody therapy (e.g., trastuzumab, pertuzumab), HER2 targeted Tyrosine Kinase inhibitors (e.g., neratinib), and/or pending breast reconstructive surgery are allowed.
* Unable to read and comprehend English (SHINE intervention currently only available in English) as indicated by being unable to complete the self-reported screening questionnaire independently

SELF-REPORTED ELIGIBILITY SCREENER EXCLUSION

* Does not have reliable access to internet (e.g., by home broadband, public network, personal data plan) by computer, tablet, smartphone etc. and is not willing to participate in the tablet lending program for this study
* Recent serious mental illness, as defined by reporting an inpatient psychiatric hospitalization within the past 12 months
* Currently participating in couple, marital, or sex therapy
* Currently pregnant (Pregnant women are excluded from this study because childbirth is accompanied by significant biological, psychological, and environmental changes that alter a woman's sexual functioning. Intervention content may not be medically appropriate for women who have recently given birth, given that medical providers commonly recommend that women avoid sexual contact for at least four to six weeks post-partum while healing.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This trial will exclusively recruit female breast cancer survivors.
Enrollment: 340 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in sexual distress as measured by the total sum score of the Female Sexual Distress Scale - Desire, Arousal, Orgasm (FSDS-DAO). The total sum score ranges from 0-60 with higher scores reflecting greater distress. | From baseline to 24 weeks
  Estimated mean change from Baseline to 24 weeks with main effect of Time will be obtained from a linear mixed models analysis of variance to account for missing data. All randomized participants will be utilized in the model (ITT analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (236):
- United States (236):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - The University of Iowa - Ankeny, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - The University of Iowa - West De Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - The University of Iowa - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - The University of Iowa - Laurel, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - CentraState Medical Center, Freehold, New Jersey
  - Hackettstown Medical Center, Hackettstown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Randolph Health Cancer Center, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Beaufort Memorial/New River Cancer Center, Okatie, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology-Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Chesapeake Regional Medical Center, Chesapeake, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Kaiser Permanente Bellevue Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be submitted to the archive 6 months post-publication and maintained according to data archive guidelines.
Access Criteria: upon request to NCORP@wakehealth.edu
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Shaffer KM, Reese JB, Dressler EV, Glazer JV, Cohn W, Showalter SL, Clayton AH, Danhauer SC, Loch M, Kadi M, Smith C, Weaver KE, Lesser GJ, Ritterband LM. Factorial Trial to Optimize an Internet-Delivered Intervention for Sexual Health After Breast Cancer: Protocol for the WF-2202 Sexual Health and Intimacy Enhancement (SHINE) Trial. JMIR Res Protoc. 2024 Aug 19;13:e57781. doi: 10.2196/57781. PMID 39159450